CLINICAL TRIAL: NCT06428032
Title: Functional and Neuroplastic Effects of Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) in Children With Bilateral Cerebral Palsy: a Randomized Controlled Trial
Brief Title: Functional and Neuroplastic Effects of HABIT-ILE in Children With Bilateral Cerebral Palsy
Acronym: FuN HABIT-ILE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Responsible Party: Principal Investigator, Rodrigo Araneda, PhD, Principal Investigator, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEUROLAB_UNAB_001
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
Keywords: HABIT-ILE; Intensive motor therapy; Motor skill learning; Children
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double period (Experimental): Subjects will receive 130 hours of HABIT-ILE performed in two intervention periods as camp format for 6,5-hours/day, 5 days/week for two weeks. Each intervention period will be 6-months apart.
  Interventions: Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities
- Single period (Experimental): Subjects will receive 65 hours of HABIT-ILE performed in one intervention period as camp format for 6,5-hours/day, 5 days/week for two weeks
  Interventions: Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities

INTERVENTIONS:
Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities — Structured bimanual tasks training, with gradual increase in motor difficulty, requiring increased postural adjustments and the use of the lower extremities.
  Other Names: HABIT-ILE
  Arms: Double period
Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities — Structured bimanual tasks training, with gradual increase in motor difficulty, requiring increased postural adjustments and the use of the lower extremities.
  Other Names: HABIT-ILE
  Arms: Single period

SUMMARY:
This randomized controlled trial will compare the effects of neuroplastic and functional changes of Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) when presented in two periods (2HG; n=24) versus a single period (1HG; n=24) in people with bilateral CP. The 1HG will receive 65 hours of HABIT-ILE over one intervention period; the 2HG will receive 130 hours over two intervention periods, within 6 months apart. Children will be assessed at 6 time points: baseline, three weeks after the start, at 3, 6, 7 and 9 months after the start of the study.

DETAILED DESCRIPTION:
This study aims to compare, for the first time, the effects of a double period of HABIT-ILE therapy on functional and neuroplastic changes against a single period, in people with bilateral cerebral palsy (CP). Previous HABIT-ILE protocols have only assessed the effects of a single intervention period. Still, the literature suggests a possible dose-response relationship between the number of intensive therapy periods and progress in motor function.

A randomized controlled trial will be conducted, comparing the effects of a double period of HABIT-ILE; (2HG; n=24) versus a single period (1HG; n=24) in children and youth with bilateral CP. Each HABIT-ILE period will consider 6.5 hours of intervention during 10 consecutive working days. Children will be assessed at 6-time points: baseline, three weeks after, at 3 months, at 6 months, at 7 months, and at 9 months, to evaluate the long-term effect of HABIT-ILE and the summative effects of the double period in functional and neuroplastic variables. The 1HG will receive only 65 hours of HABIT-ILE after baseline; the 2HG will perform 130 hours over two intervention periods, after baseline and again at 6 months.

Overall, this study aims to provide evidence for the effectiveness of HABIT-ILE in producing functional and neuroplastic changes in children with bilateral CP. It will allow us to approach the possible mechanisms underlying the effect of HABIT-ILE.

ELIGIBILITY:
Inclusion Criteria:

* Children with medical diagnosis of bilateral cerebral palsy
* Cognitive capacity and language that allows understanding and following the therapist's instructions.
* Manual Ability Classification System (MACS) levels I to III
* Bimanual Fine Motor Function (BFMF) levels I to III
* Gross Motor Function Classification System (GMFCS) levels I to III

Exclusion Criteria:

* Severe visual problems
* Movement restriction due to orthopedic surgery in less than a year
* Treatment with botulinum toxin and/or baclofen pump in the last 6 months
* Contraindications to receive transcranial magnetic stimulation (epileptic history, metallic implants, neoplasm, etc.)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Gross Motor Function | Baseline (T0), two weeks after start (T1), at 3 months (T2), at 6 months (T3), at 7 months (T4), and at 9 months (T5)
  The Gross Motor Function Measure is a standardized observational instrument designed to measure changes in gross motor function over time or following an intervention in children and youth with cerebral palsy using Rasch analysis. It is scored on a scale of 0 to 3, where 0 means the person cannot perform the activity and 3 means the person can complete the item. The score is converted to a percentage. A higher percentage means a better gross motor function.

SECONDARY OUTCOMES:
Both Hands Assessment (BoHA) | Time Frame: Baseline (T0), two weeks after start (T1), at 3 months (T2), at 6 months (T3), at 7 months (T4), and at 9 months (T5)]
  The Both Hands Assessment is a valid test for children with mild to moderate bilateral manual abilities impairments. It can evaluate bimanual activity performance and the level of upper extremity asymmetry. It rates performance between 1 (does not do) and 4 (effective). The final score is converted to BoHA units (logit 0 - 100), where higher scores reflect better bimanual use.
Melbourne 2 Assessment (MA2) | Time Frame: Baseline (T0), two weeks after start (T1), at 3 months (T2), at 6 months (T3), at 7 months (T4), and at 9 months (T5)]
  The Melbourne 2 Assessment (MA2) assesses the unilateral performance of the upper extremities, quantifying the dexterity, fluency, accuracy, and range of movement during several tasks of reaching and manipulation. The result is obtained as a percentage of the function of each item. A higher percentage means a better unilateral performance of the upper extremity.
Test of Arm Selective Control (TASC) | Time Frame: Baseline (T0), two weeks after start (T1), at 3 months (T2), at 6 months (T3), at 7 months (T4), and at 9 months (T5)
  The TASC test assesses the selective voluntary motor control of upper limbs in individuals with cerebral palsy. The participant must execute eight movements in the upper extremity. The execution of each sequence will be assessed on a scale of 0, 1, or 2, from absence, impairment, or normality of voluntary selective motor control, respectively, with a maximum of 16 points per side and 32 points overall.
Selective Control Assessment of the Lower Extremity (SCALE) | Time Frame: Baseline (T0), two weeks after start (T1), at 3 months (T2), at 6 months (T3), at 7 months (T4), and at 9 months (T5)
  The SCALE test assesses the selective voluntary motor control of lower limbs in individuals with cerebral palsy. The participant must execute five movements in the lower extremity. The execution of each sequence will be assessed on a scale of 0, 1 or 2, from absence, impairment, or normality of voluntary selective motor control respectively, with a maximum of 10 points per side and 20 points overall.
Six minutes walk test (6MWT) | Time Frame: Baseline (T0), two weeks after start (T1), at 3 months (T2), at 6 months (T3), at 7 months (T4), and at 9 months (T5)
  The 6MWT measures the maximum distance a participant can walk in a 6-minute period in a 30-meter corridor at his or her own pace. More distance walked (in meters) indicates better performance.
Attention network test (ANT) | Time Frame: Baseline (T0), two weeks after start (T1), at 3 months (T2), at 6 months (T3), at 7 months (T4), and at 9 months (T5)
  The ANT assesses the efficiency of the three attentional networks: alerting, orienting, and executive control networks. It measures the accuracy (in terms of the amount of errors) and the reaction time (milliseconds) of each network. Fewer errors mean more accuracy, the lower the score, the faster the reaction time.
ABILHAND-Kids questionnaire | Time Frame: Baseline (T0), two weeks after start (T1), at 3 months (T2), at 6 months (T3), at 7 months (T4), and at 9 months (T5)
  This parent's filled questionnaire measures the ability of the participant with cerebral palsy to perform activities of daily living that require the use of the upper extremities. The difficulty to perform the activities are rating as "Impossible", "Difficult" or "Easy". The result is obtained in logits and can be interpreted as a percentage, where 0% indicates minimum ability and 100% maximum ability to perform the activities.
ACTIVLIM-CP questionnaire | Time Frame: Baseline (T0), two weeks after start (T1), at 3 months (T2), at 6 months (T3), at 7 months (T4), and at 9 months (T5)
  This parent's filled questionnaire measures a child performance of daily activities requiring the use of the upper and/or the lower extremities through 43 items specific to patients with cerebral palsy. It ranges from - 7 to +7 logits (higher score means better performance). The result is obtained in logits and can be interpreted as a percentage, where 0% indicates minimum ability and 100% maximum ability to perform the activities.
Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) | Time Frame: Baseline (T0), two weeks after start (T1), at 3 months (T2), at 6 months (T3), at 7 months (T4), and at 9 months (T5)
  This parent's filled questionnaire measures the performance of the child in the daily life activities and movement domains, focusing on the capacity of upper extremities and lower extremities during these activities. It ranges from 20 to 80 (higher score means better performance).
Participation and Environment Measure - Children and Youth (PEM-CY) | Time Frame: Baseline (T0), two weeks after start (T1), at 3 months (T2), at 6 months (T3), at 7 months (T4), and at 9 months (T5)
  This parent's filled questionnaire measures participation of children and youth with or without disability, in the home, school and community, along with environmental factors within each of these settings. For each environment, it assesses how frequently they participate in a given activity (8-point scale; 0-7), how involved they are in that activity (5-point scale; 1-5), and whether they want to make a change in the type of participation they perform (6-point scale; 1-6). For each setting, the participation frequency (percentage), involvement (score 1-5), desires for change (percentage), and environmental supportiveness (percentage) are calculated.
Canadian Occupational Performance Measure (COPM) | Time Frame: Baseline (T0), two weeks after start (T1), at 3 months (T2), at 6 months (T3), at 7 months (T4), and at 9 months (T5)
  This is an interview-setting designed to capture a patient's self-perception of performance and satisfaction of it in everyday activities, observed over time. During the interview, parents set up 5 activities considered difficult in daily life. These are then assessed, in a 1 to 10 scale, regarding the child's self-perception of performance and satisfaction of it. The total score is the average of the scores for perception and satisfaction separately (score from 1 to 10; higher score means better performance/satisfaction).
Behaviour Rating Inventory of Executive Function (BRIEF-2) | Time Frame: Baseline (T0), at 3 months (T2), at 6 months (T3), and at 9 months (T5)
  The BRIEF-2 is a caregiver-reported questionnaire measuring executive functioning in children between 5 and 18 years old. It consists of 63 items arranged in nine scales: inhibition, self-monitoring, flexibility, emotional control, initiative, working memory, planning and organization, task supervision, and organization of materials. It is scored using T scores (Range= 34 - 90; Mean=50, Standard Deviation=10), where higher scores indicate greater problems with executive functioning.
Changes of peak-to-peak amplitude of motor evoked potential | Time Frame: Baseline (T0), two weeks after start (T1), at 6 months (T3), and at 7 months (T4)
  A single-pulse transcranial magnetic stimulation is a noninvasive technique that directly assesses cortical function and connectivity in the motor system. It will be used to assess the corticospinal tract excitability in both brain hemispheres. It will stimulate the primary motor cortex with a figure-8 coil, searching for the first dorsal interosseous muscle area. The changes of peak-to-peak amplitude of motor evoked potential will be measured in milliAmpere (mA).
Changes of Resting Motor Threshold | Time Frame: Baseline (T0), two weeks after start (T1), at 6 months (T3), and at 7 months (T4)
  A single-pulse transcranial magnetic stimulation is a noninvasive technique that directly assesses cortical function and connectivity in the motor system. It will be used to assess the corticospinal tract excitability in both brain hemispheres. It will stimulate the primary motor cortex with a figure-8 coil, searching for the first dorsal interosseous muscle area. The changes of resting motor threshold will be measured in percentage.
Changes of latency in motor evoked potential | Time Frame: Baseline (T0), two weeks after start (T1), at 6 months (T3), and at 7 months (T4)
  A single-pulse transcranial magnetic stimulation is a noninvasive technique that directly assesses cortical function and connectivity in the motor system. It will be used to assess the corticospinal tract excitability in both brain hemispheres. It will stimulate the primary motor cortex with a figure-8 coil, searching for the first dorsal interosseous muscle area. The changes of latency in motor evoked potential will be measured in milliseconds.
Changes of oxyhemoglobin concentration in sensorimotor cortex | Time Frame: Baseline (T0), two weeks after start (T1), at 6 months (T3), and at 7 months (T4)
  A functional near-infrared spectroscopy will be used to assess cortical activity. It is a noninvasive brain imaging tool that records optical density measurements to determine the change in oxyhemoglobin concentration (μM) in sensorimotor cortex area during manual tasks.
Changes of oxyhemoglobin concentration in prefrontal cortex | Time Frame: Baseline (T0), two weeks after start (T1), at 6 months (T3), and at 7 months (T4)
  A functional near-infrared spectroscopy will be used to assess cortical activity. It is a noninvasive brain imaging tool that records optical density measurements to determine the change in oxyhemoglobin concentration (μM) in prefrontal cortex area during manual tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Araneda, PhD, Principal Investigator — Universidad Nacional Andres Bello
Locations (1):
- Exercise and Rehabilitation Sciences Institute, Universidad Nacional Andres Bello, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No